CLINICAL TRIAL: NCT00651443
Title: A Phase I, Open Label Study to Evaluate the Mechanism of Action of Galiximab in Subjects With Previously Untreated Follicular Non-Hodgkin's Lymphoma
Brief Title: Mechanism of Action of Galiximab in Subjects With Previously Untreated Follicular Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A company's strategic decision to focus on areas whereit believes it can be competitive and decided to exit Oncology
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114-NH-103
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Lymphoma, Non-Hodgkin's
Keywords: galiximab; Untreated NHL; antibody; open-label
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — galiximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Galiximab

INTERVENTIONS:
Drug: Galiximab — Galiximab 500 mg/m2 IV once weekly times 4, followed by Galiximab 500 mg/m2 IV once monthly times 4 as an extended dosing regimen.

SUMMARY:
The purpose of the study is to evaluate the mechanism(s) of action of galiximab in subjects with previously untreated follicular NHL.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (signed and dated).
* Age equal or greater than 18 at the time of consent.
* Histologically confirmed follicular NHL according to the Revised European American Lymphoma (REAL)/ World Health Organization (WHO) classification (from initial diagnosis) Grades 1,2, or 3a.
* At least 2 malignant lymph nodes of similar size (>1 cm in minimal dimension) and location that are readily accessible for excisional biopsy at the time of study entry.
* Consent to 1 pretreatment and 1 post-treatment excisional biopsy of accessible tumor.
* Acceptable hematologic, hepatic, and renal function parameters.
* WHO Performance Status equal or less than 2.
* Subjects of reproductive potential must agree to follow accepted birth control methods.

Exclusion Criteria:

* Presence of lymphoma in CNS.
* Previous systemic anticancer treatment for NHL (including but not limited to radiation, myeloablative, or investigational therapy).
* Concurrent treatment with systemic steroids within 14 days of Day 1.
* Evidence of transformed lymphoma.
* Presence of malignancies within 3 years of Study Day 1 (except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of breast, or basal or squamous cell skin cancer).
* History of HIV infection or AIDS.
* Serious nonmalignant disease.
* Pregnant.
* Inability to comply with study and follow-up procedures.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Mechanism of action of galiximab given as a single agent in previously untreated subjects with follicular NHL. | 24 months

SECONDARY OUTCOMES:
1) Safety and tolerability of Galiximab when administered as a single agent in an extended dosing regimen in previously untreated subjects with follicular NHL. 2) Evaluation of preliminary clinical activity of galiximab. | 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Buffalo, New York, United States